CLINICAL TRIAL: NCT02230540
Title: Intermittent Catheterization in Spinal Cord Injured Men
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP250
Record Dates: First submitted 2014-08-28; First posted 2014-09-03 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-02

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence A (Experimental): Catheterization with SelfCath (comparator) followed by measurement of residual urine.
  Then catheterization with Product A in different positions. Measurement of residual urine at different positions.
  Interventions: Device: SelfCath (comparator); Device: Product A SelfCath and urine bag, Conveen Security+
- Sequence B (Experimental): Based on results from sequence A, sequence B may or may not be initiated.
  Catheterization with SelfCath (comparator) followed by measurement of residual urine.
  Then catheterization with Product B in different positions. Measurement of residual urine at different positions.
  Interventions: Device: SelfCath (comparator); Device: Product B SelfCath and urine bag, Conveen Contour

INTERVENTIONS:
Device: SelfCath (comparator) — Commercially available CE-marked catheter for urinary drainage.
Device: Product A SelfCath and urine bag, Conveen Security+ — SelfCath and urine bag, Conveen Security+ (both commercially available CE-marked devices).
  Arms: Sequence A
Device: Product B SelfCath and urine bag, Conveen Contour — SelfCath and urine bag, Conveen Contour (both commercially available CE-marked devices).
  Arms: Sequence B

SUMMARY:
The aim of this investigation is to study how the position of different catheters affect drainage of the bladder.

ELIGIBILITY:
Inclusion Criteria:

* Has given written informed consent
* Is at least 18 years of age and has full legal capacity
* Is a male
* Has an Spinal Cord Injury diagnosis

Exclusion Criteria:

* Participating in other interventional clinical investigations or have previously participated in this investigation
* Known hypersensitivity toward any of the test products
* Serious abdominal scars
* Symptoms of urinary tract infections

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per Bagi, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Per Bagi, Copenhagen, Denmark

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence A: Catheterization with SelfCath (comparator) followed by measurement of residual urine.
  Then catheterization with Product A in different positions. Measurement of residual urine at different positions.
  SelfCath (comparator): Commercially available CE-marked catheter for urinary drainage.
  Product A SelfCath and urine bag, Conveen Security+: SelfCath and urine bag, Conveen Security+ (both commercially available CE-marked devices).
- Sequence B: Based on results from sequence A, sequence B may or may not be initiated.
  Catheterization with SelfCath (comparator) followed by measurement of residual urine.
  Then catheterization with Product B in different positions. Measurement of residual urine at different positions.
  SelfCath (comparator): Commercially available CE-marked catheter for urinary drainage.
  Product B SelfCath and urine bag, Conveen Contour: SelfCath and urine bag, Conveen Contour (both commercially available CE-marked devices).
Period: Overall Study
Arm/Group | Sequence A | Sequence B
Started | 8 | 0 (The study was terminated before initiation of sequence B. Sequence B was therefore not initiated.)
Completed | 8 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequence A: Catheterization with SelfCath (comparator) followed by measurement of residual urine.
  Then catheterization with Product A in different positions and measurement of residual urine.
  SelfCath (comparator): Catheter for urinary drainage.
  Product A: SelfCath and urine bag, Conveen Security+ (both commercially available CE-marked devices).
Arm/Group | Sequence A
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Region of Enrollment [Number; unit: participants]
  Denmark | 8

OUTCOME MEASURES:

1. Primary Outcome: Residual Volume Less Than 100ml
Description: The primary endpoint was "Residual volume less than 100 ml (Yes/No)" assessed after catheterization when placed at fixed heights (25, 20, 15, 10 and 0 cm) over the wheelchair seat.
  Prior to the catheterization corresponding to height 25 cm, a solution was instilled into the bladder to ensure a volume equal to 300 ml. The residual volume at height 25 cm was then calculated as 300 ml minus the volume emptied during catheterization. The residual volume corresponding to height 20 cm was calculated as the residual volume corresponding to height 25 minus the additional volume emptied at height 20. The residual volume corresponding to height 15, 10 and 0 cm were derived similarly.
  Calculated residual volumes were negative, likely due to faulty ultrasound scans performed on subjects in sitting position. Consequently, the changes in bladder volumes, re-worded from "300ml - collected volume <100ml" to "collected volume > 200ml", were used to interpret the primary endpoint.
Time Frame: 2-4 hours
Measure: Number; unit: Subjects with successful catheterization
Arm/Group | Sequence A
Number analyzed (Participants) | 8
Subjects with successful catheterization
  Height 25cm | 6
  Height 20cm | 6
  Height 15cm | 6
  Height 10cm | 6
  Height 0cm | 7

ADVERSE EVENTS:
Arm/Group | Sequence A
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators who want to publish/present results based on own data from a Coloplast-sponsored investigation, must send the publication/presentation to sponsor for review 60 days prior to submission. Sponsor reserves the right to delay publications to avoid compromising intellectual property. Publications of sub-analyses may be delayed by sponsor until main results of investigation have been published.